CLINICAL TRIAL: NCT05856747
Title: An Open-Label, Single-Center, Single-Period Study to Compare Two Bioanalytical Assays for Tebipenem Following Administration of Oral Tebipenem Pivoxil Hydrobromide in Healthy Adult Volunteers
Brief Title: A Study to Compare Two Bioanalytical Assays for Tebipenem
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Spero Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPR994-109
Record Dates: First submitted 2023-05-03; First posted 2023-05-12 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2023-07

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — tebipenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- TBP-PI-HBr 600 mg (Experimental): Healthy participants meeting eligibility criteria will receive a single oral dose of TBP-PI-HBr 600 mg tablets (2 x 300 mg) on Day 1 under fasted conditions.
  Interventions: Drug: TBP-PI-HBr

INTERVENTIONS:
Drug: TBP-PI-HBr — TBP-PI-HBr tablets.
  Other Names: SPR994

SUMMARY:
The primary purpose of the study is to compare the concentrations of tebipenem (TBP), the active moiety of tebipenem pivoxil hydrobromide (TBP-PI-HBr), as determined by two bioanalytical assays, a whole blood assay and a plasma assay, following a single oral dose of TBP-PI-HBr 600 milligram (mg) tablets in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ≥18.0 and ≤32.0 kilograms per meter square (kg/m^2) at Screening visit.
* Medically healthy with no clinically significant medical history, abnormalities in physical examination, laboratory variables, vital signs or electrocardiogram (ECG) at the time of Screening visit and Check-in (Day-1), as deemed by the investigator or designee.
* Have suitable venous access for repeated blood sampling.

Exclusion Criteria:

* Any clinically significant medical history or observations at the time of Screening visit or Check-in (Day -1) not specifically excluded in other criteria that, in the opinion of the investigator or designee, may confound the results of the study, compromise the safety of the participant or otherwise render the participant unsuitable for participation.
* Use/receipt of any prescription or non-prescription medication, herbal products, vitamins or vaccines within 14 days (or 5 half-lives whichever is longer) prior to Check-in (Day -1).
* Positive coronavirus disease (COVID-19) screening test using polymerase chain reaction (PCR) or antigen assay at Screening visit or Check-in (Day -1).
* Donation or significant blood loss of more than 500 milliliter (mL) of blood within 56 days prior to enrollment, or receipt of a blood transfusion within 1 year prior to enrollment; plasma donation within 7 days prior to dosing.
* ECG with corrected QT interval by Fridericia (QTcF) interval duration equal or greater than 450 milliseconds (msec) for males and 470 msec for females obtained after at least 5 minutes in a supine or semi-recumbent position at quiet rest at Screening visit or Check-in (Day -1).

Other inclusion and exclusion criteria as per protocol may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-05-04 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Percentage of Tebipenem (TBP) Samples With Converted (From Whole Blood Measurements) and Measured Plasma Concentrations That Have a Difference not Exceeding ±20% of the Mean of the Concentrations | Pre dose and at multiple time points post dose on Day 1
Area Under the Plasma Concentration-time Curve Extrapolated to Infinity (AUC0-∞) of TBP | Pre dose and at multiple time points post dose on Day 1
Maximum Plasma Concentration (Cmax) of TBP | Pre dose and at multiple time points post dose on Day 1

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) | From first dose of study drug up to Day 6

CONTACTS AND LOCATIONS:
Locations (1):
- BioPharma Services, Creve Coeur, Missouri, United States

IPD SHARING:
Plan to Share IPD: No